CLINICAL TRIAL: NCT02122159
Title: A Phase I/II, Open-Label, Prospective Study to Determine the Safety and Tolerability of Sub-retinal Transplantation of Human Embryonic Stem Cell Derived Retinal Pigmented Epithelial (MA09-hRPE) Cells in Patients With Geographic Atrophy Secondary to Myopic Macular Degeneration
Brief Title: Research With Retinal Cells Derived From Stem Cells for Myopic Macular Degeneration
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study to be revised. Future plans to be determined.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Ocata Therapeutics (Industry)
Responsible Party: Principal Investigator, Steven Schwartz, Chief, Retina Division, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSEI MA09-hRPE MMD
Record Dates: First submitted 2014-04-01; First posted 2014-04-24 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Myopic Macular Degeneration
Keywords: safety; tolerability; RPE cellular therapy; MMD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MA09-hRPE Cellular Therapy (Experimental): MA09-hRPE cells for transplantation will be provided by Ocata Therapeutics as a suspension frozen to the temperature of liquid nitrogen (approximately -196 °C). They will be processed at UCLA under GMPs according to protocol. Following vitrectomy performed under general anesthesia or waking sedation at the surgeon's discretion, hRPE cells will be introduced into a subretinal bleb formed by the injection of balanced salt solution (BSS). Direct viewing will guide the implantation of thawed and washed MA09-hRPE cells, resuspended in BSS, into the created bleb over a period of one minute. To avoid cell reflux, the cannula used to introduce the cells will be held in position for an additional minute. A suspension of either 50,000 MA09-hRPE cells (first cohort), 100,000 MA09-hRPE cells (second cohort), 150,000 MA09-hRPE cells (third cohort) or 200,000 MA09-hRPE cells (fourth cohort) in 150 uL of BSS plus will be implanted over 1 minute in the space created.
  Interventions: Biological: MA09-hRPE Cellular Therapy

INTERVENTIONS:
Biological: MA09-hRPE Cellular Therapy — A suspension of either 50,000 MA09-hRPE cells (first cohort), 100,000 MA09-hRPE cells (second cohort), 150,000 MA09-hRPE cells (third cohort) or 200,000 MA09-hRPE cells (fourth cohort) in 150 uL of BSS plus will be implanted over 1 minute in the space created.

SUMMARY:
Pathologic myopia is a major cause of legal blindness worldwide. In myopic macular degeneration (MMD), there is degeneration of the retinal pigment epithelial (RPE) layer, and associated photoreceptors, resulting in vision loss. There is currently no standard treatment for MMD.

Transplantation of intact sheets of RPE and suspensions of isolated individual RPE cells as well as autologous translocation of RPE cells has been attempted as treatment for AMD. Human photoreceptors are comprised of two cell types-rods and cones. Both have a close relationship with the outermost retinal cells, the retinal pigmented epithelium (RPE). The RPE is located between the choroid and the photoreceptors. The RPE maintains photoreceptor function by recycling photopigments,delivering, metabolizing and storing vitamin A, phagocytosing rod photoreceptor outer segments, transporting iron and small molecules between retina and choroid, maintaining Bruch's membrane and absorbing stray light to allow better image resolution. In essence, the RPE layer is critical to the function and health of photoreceptors and the retina as a whole.

Human PRE (hRPE) transplantation may be a viable option for treatment of degenerative diseases of the retina.

MA09-hRPE cells are fully differentiated human RPE cells derived from embryonic stem cells. Transplanted hRPE cells prepared by Advanced Cell Technology have been studied in rodent models of macular degenerative disease. The data suggests that the subretinal injection of ACT's hRPE cell products rescues, or at least delays, loss of visual function in two animal models of retinal degenerative diseases.

The main purpose of this study is to evaluate the safety and tolerability of MA09-hRPE cellular therapy in patients with Myopic Macular Degeneration (MMD). Another objective is to evaluate potential efficacy endpoints to be used in future studies of RPE cellular therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female over 40 years of age.
* Patient should be in sufficiently good health to reasonably expect survival for at least four years after treatment
* Axial myopia of equal to or greater than -8 diopters and/or axial length equal to or greater than 28 mm
* Clinical findings consistent with MMD with evidence of one or more areas of >250microns of geographic atrophy (as defined in the Age-Related eye Disease Study [AREDS] study) involving the central fovea.
* GA defined as attenuation or loss of RPE as observed by biomicroscopy, OCT, and FA.
* No evidence of current or prior choroidal neovascularization
* The visual acuity of the eye to receive the transplant will be no better than 20/80.
* The visual acuity of the eye that is NOT to receive the transplant will be no worse than 20/400.
* The eye with the more advanced disease and worse vision will be the study eye.
* Electrophysiological findings consistent with macula-involving geographic atrophy.
* Medically suitable to undergo vitrectomy and subretinal injection.
* Medically suitable for general anesthesia or waking sedation, if needed.
* Medically suitable for transplantation of an embryonic stem cell line:

Any laboratory value, which falls slightly outside of the normal range, will be reviewed by the Medical Monitor and Investigators to determine its clinical significance. If it is determined not to be clinically significant, the patient may be enrolled into the study.

* Normal serum chemistry (sequential multi-channel analyzer 20 [SMA-20]) and hematology (complete blood count [CBC], prothrombin time [PT], and activated partial thromboplastin time [aPTT]) screening tests. (NOTE:With the exception of abnormalities specifically identified in the exclusion criteria)
* Negative urine screen for drugs of abuse.
* Negative human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV) serologies.
* No history of malignancy (with the exception of successfully treated (excised) basal cell carcinoma[skin cancer] or successfully treated squamous cell carcinoma of the skin).
* Negative cancer screening within previous 6 months:
* complete history & physical examination;
* dermatological screening exam for malignant lesions;
* negative fecal occult blood test & negative colonoscopy within previous 7 years;
* negative chest roentgenogram (CXR);
* normal CBC & manual differential;
* negative urinalysis (U/A);
* normal thyroid exam;
* if male, normal testicular examination; digital rectal examination (DRE) and prostate specific antigen (PSA);
* if female, normal pelvic examination with Papanicolaou smear; and
* If female, normal clinical breast exam and, negative mammogram.
* If female and of childbearing potential, willing to use two effective forms of birth control during the study.
* If male, willing to use barrier and spermicidal contraception during the study.
* Willing to defer all future blood, blood component or tissue donation.
* Able to understand and willing to sign the informed consent.

Exclusion Criteria:

* Presence of active or inactive CNV.
* Presence of a posterior staphyloma.
* Presence or history of retinal dystrophy, retinitis pigmentosa, chorioretinitis, central serious choroidopathy, diabetic retinopathy or other retinal vascular or degenerative disease (i.e. AMD) other than MMD.
* History of optic neuropathy.
* Macular atrophy due to causes other than MMD.
* Presence of glaucomatous optic neuropathy in the study eye, uncontrolled IOP, or use of two or more agents to control IOP (acetazolamide, beta blocker, alpha-1-agonist, antprostaglandins, carbonic anhydrase inhibitors).
* Cataract of sufficient severity likely to necessitate surgical extraction within 1 year.
* History of retinal detachment repair in the study eye.
* History of malignancy (with the exception of successfully treated [excised] basal cell carcinoma [skin cancer] or successfully treated squamous cell carcinoma of the skin).
* History of myocardial infarction in previous 12 months.
* History of cognitive impairments or dementia which may impact the patients ability participate in the informed consent process and to appropriately complete evaluations.
* Any immunodeficiency.
* Any current immunosuppressive therapy other than intermittent or low dose corticosteroids.
* Alanine transaminase/aspartate aminotransferase (ALT/AST) >1.5 times the upper limit of normal or any known liver disease.
* Renal insufficiency, as defined by creatinine level >1.3 mg/dL.
* A hemoglobin concentration of less than 10gm/dL, a platelet count of less than 100k/mm3 or an absolute neutrophil count of less than 1000/mm3 at study entry.
* Serologic evidence of infection with Hepatitis B, Hepatitis C, or HIV.
* Current participation in any other clinical trial.
* Participation within previous 6 months in any clinical trial of a drug by ocular or systemic administration.
* Any other sight-threatening ocular disease.
* Any history of retinal vascular disease (compromised blood-retinal barrier.
* Glaucoma.
* Uveitis or other intraocular inflammatory disease.
* Significant lens opacities or other media opacity.
* Ocular lens removal within previous 3 months.
* Ocular surgery in the study eye in the previous 3 months
* If female, pregnancy or lactation.
* Any other medical condition, which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromises patient safety, or interferes with the interpretation of the study results.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety of hESC-derived RPE cells | 12 months
  The transplantation of hESC-derived RPE cells MA09-hRPE will be considered safe and tolerated in the absence of:
  * Any grade 2 (NCI grading system) or greater adverse event related to the cell product
  * Any evidence that the cells are contaminated with an infectious agent
  * Any evidence that the cells show tumorigenic potential

SECONDARY OUTCOMES:
Evidence of successful engraftment | 12 months
  Evidence of successful engraftment will consist of:
  * Structural evidence (OCT imaging, fluorescein angiography, slit-lamp examination with fundus photography) that cells have been implanted in the correct location
  * Electroretinographic evidence (mfERG) showing enhanced activity in the implant location
Evidence of rejection | 12 months
  Evidence of rejection will consist of:
  • Structural (imaging) evidence that implanted MA09-hRPE cells are no longer in the correct location or the presence of vascular leakage
  If enhanced electroretinographic activity is observed after the transplantation, subsequent electroretinographic evidence that activity has returned to pre-transplant conditions may be an indication of graft rejection

CONTACTS AND LOCATIONS:
Overall Officials: Steven Schwartz, MD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No